CLINICAL TRIAL: NCT05709951
Title: Effects of Functional Versus Core Stability Exercises on Pain and Sleep Quality in Patients With Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RiphahIU fatimatariq1
Record Dates: First submitted 2023-01-04; First posted 2023-02-02 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Primary Dysmenorrhea
Keywords: Core stability,Exercises,Primary dysmenorrhea,sleep quality
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Who Masked: Participant
Masking Description: Blinding
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional exercises (Active Comparator): Piriformis stretching Cobra pose Sit up Bridging exercise
  Interventions: Other: Functional Exercises
- Core Stability Exercises (Active Comparator): Pelvic bridging Plank Cat and camel Curl up
  Interventions: Other: Core Stability Exercises

INTERVENTIONS:
Other: Functional Exercises — The patients were requested to perform these functional exercises for 4 days per week three times for 20 min (8 weeks).
  Other Names: Exercises
  Arms: Functional exercises
Other: Core Stability Exercises — The patients were requested to perform 4 core strengthening exercises for 4 days per week three times for 20 min (8 weeks)
  Other Names: Exercises
  Arms: Core Stability Exercises

SUMMARY:
To compare the effects of Functional and Core stability exercises on pain and sleep quality in Patients with Primary Dysmenorrhea and to check the results of exercises may be effective in pain during Menstrual and before cramping in menses.

ELIGIBILITY:
Inclusion Criteria:

* Having used medication for menstrual pain and not having used oral contraceptives during the three months prior to admission to the study.
* Pain must be periodic (at least following 3 menstrual cycles).
* Lower abdominal cramps pain ends after periods and gradually diminish over 12 to 72 hrs.
* No history of blood disorders including thalassemia and folate or iron-deficiency anemia

Exclusion Criteria:

* Pelvic inflammatory disease
* Ovarian cysts
* Chronic abdominal pain
* Fibroids, obstructive endometrial polyps,
* Irritable bowel syndrome
* Major abdominal or pelvic surgery
* Intrauterine devices.

Ages: 15 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — Female with primary dysmenorrhea
Enrollment: 24 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2023-02 (Estimated); Study Completion 2023-02 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale for lower abdominal pain | 8 week
  The subjective and verified visual analogue scale is used to quantify both acute and chronic pain (1). On the 10 cm line, scores are recorded by making a mark. Pain intensity is measured along a 10-cm line with 0 denoting "no pain" and 10 denoting "worst pain."
Menstrual Symptom Questionnaire | 8 weeks
  Menstrual Symptom Questionnaire (MSQ) to assess dysmenorrhea symptoms. The MSQ is a 24 item self-report measure which assesses menstrual pain and symptoms (e.g. 'I have cramps that begin on the first day of my period'; 'I feel depressed for several days before my period'). The score on each item ranges from 1 (never) to 5 (always) with a higher composite score indicating more symptoms.
Pittsburgh Sleep Quality Index | 8 week
  Pittsburgh Sleep Quality Index (PSQI) evaluates sleep disruptions and quality over a 1-month period. In scoring the PSQI, seven component scores are derived, each scored 0 (no difficulty) to 3 (severe difficulty).

CONTACTS AND LOCATIONS:
Overall Officials: Fatima Tariq, PhD, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No